CLINICAL TRIAL: NCT04601935
Title: A Single-center Exploratory Clinical Study to Evaluate the Safety, Tolerability, and Efficacy of a BCMA-targeted Universal LCAR-BCX Cells in Patients With Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Weijun Fu (Other)
Collaborators: Nanjing Legend Biotech Co. (Industry)
Responsible Party: Sponsor-Investigator, Weijun Fu, Director of Hematology Department, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BM2L202004
Record Dates: First submitted 2020-10-09; First posted 2020-10-26 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Relapsed/Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- LCAR-BCX cells product (Experimental): Each subject will be given a single-dose infusion in each dose levelThe dose-finding phase of this study is designed primarily using the Bayesian optimal interval (BOIN) method, which is combined with accelerated titration at the beginning of the study to assess incidence of DLT (dose-limiting toxicity) and estimate MTD (maximum tolerated dose).
  Interventions: Biological: LCAR-BCX cells product

INTERVENTIONS:
Biological: LCAR-BCX cells product — In this study, LCAR-BCX CAR+ cells will be evaluated at 5 dose levels including 0.25 × 10^6 cells/kg, 0.5 × 10^6 cells/kg, 1.0 × 10^6 cells/kg, 2.0 × 10^6 cells/kg, and 4.0 × 10^6 cells/kg, with 0.25 × 10^6 cells/kg as the starting dose, to determine RP2D for LCAR-BCX cell therapy

SUMMARY:
This is a prospective, single-arm, single-center, open-label dose-finding and dose-expansion study that evaluates the safety, tolerability, PK, and anti-tumor efficacy of LCAR-BCX cells in subjects with relapsed/refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to participate in the clinical study; fully understands and informed the study contents, and signs the informed consent form.
* Chinese subjects ≥ 18 years of age.
* Documented initial diagnosis of MM according to IMWG diagnostic criteria.
* Presence of measurable disease at screening.
* Received a PI and an IMiD (except thalidomide).
* Received at least 3 prior lines of therapy for multiple myeloma, undergone at least 1 complete cycle of treatment for each line, unless progressive disease (PD) was documented by IMWG criteria as the best response to the regimen. Also, subjects refractory or intolerant to any PI and any IMiD in their previous treatment afterwards are eligible.
* Expected survival ≥ 3 months.

Exclusion Criteria:

* No response to prior BCMA-targeted CAR-T therapy (except for subjects who relapsed after CR to prior CAR-T therapy).
* Prior treatment with any BCMA-targeted monoclonal antibody.
* Diagnosed or previously treated for other invasive malignancies other than multiple myeloma, with the following exceptions:

  * Malignancies treated with curative intent and with no known active disease present for ≥ 2 years before enrollment; or
  * Adequately treated non-melanoma skin cancer without current evidence of disease.
* Prior anti-tumor therapies as follows (prior to conditioning):

  * Monoclonal antibody treatment for multiple myeloma within 21 days
  * Targeted therapy, epigenetic therapy, or treatment with an investigational product, or used an invasive investigational medical device within 14 days or at least 5 half-lives (whichever is less)
  * Cytotoxic therapy within 14 days
  * Proteasome inhibitor therapy within 14 days
  * Radiotherapy within 14 days. However, if the radiation field covers ≤ 5% of bone marrow reserve, the subject is eligible to participate in the study regardless of the end date of radiaotherapy
  * Immunomodulatory agent therapy within 7 days.
* Toxicities (excluding hematology and chemistry indicators specified in the inclusion criteria) associated with prior anti-tumor therapy must have recovered to baseline level or to ≤ Grade 1 except for alopecia or peripheral neuropathy.
* Occurrence of the following cardiac disorders:

  * NYHA stage III or IV congestive heart failure
  * Myocardial infarction or coronary artery bypass graft (CABG) ≤ 6 months prior to enrollment
  * History of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration
  * History of severe non-ischemic cardiomyopathy
  * Impaired cardiac function (LVEF < 45%) as assessed by echocardiography or multi-gated acquisition (MUGA) scan (performed ≤ 8 weeks prior to screening).
* Received either of the following treatments:

  * An allogeneic stem cell transplantation for multiple myeloma
  * An autologous stem cell transplantation ≤ 16 weeks prior to infusion.
* Known active, or prior history of, central nervous system (CNS) involvement or clinical signs of meningeal involvement of multiple myeloma.
* Supplemental oxygen required to maintain adequate oxygen saturation (≥ 95%).
* Uncontrolled diabetes.
* Stroke or epilepsy seizure within 6 months prior to signing ICF (except for old lacunar infarction).
* Plasma cell leukemia (plasma cells > 2.0 × 109/L per standard differential), Waldenström's macroglobulinemia, POEMS syndrome, or primary AL amyloidosis at the time of screening.
* Seropositive for human immunodeficiency virus (HIV).
* Positive for any one of hepatitis B surface antigen (HBsAg), hepatitis B virus deoxyribonucleic acid (HBV DNA), hepatitis C antibody (HCV-Ab), hepatitis C virus ribonucleic acid (HCV RNA), or human immunodeficiency virus antibody (HIV-Ab).
* Vaccinated with live, attenuated vaccine within 4 weeks prior to screening.
* Known life-threatening allergies, hypersensitivity, or intolerance to CAR-T cells or its excipients, including DMSO.
* Serious underlying medical condition, such as:

  * Evidence of serious active viral, bacterial, or uncontrolled systemic fungal infection
  * Active autoimmune disease or a history of autoimmune disease within 3 years
  * Overt clinical evidence of dementia or altered mental status
  * Any history of Parkinson's disease or other neurodegenerative disorder.
* Any issue that would impair the ability of the subject to receive or tolerate the planned treatment at the investigational site, to understand the informed consent, or any condition that, in the opinion of the investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being), or any condition that may prevent, limit, or confound protocol-specified assessments.
* Male subjects who plan to father a child while enrolled in the study or within 1 year after receiving study treatment.
* Female subjects who are pregnant, breastfeeding, or plan to become pregnant while enrolled in the study or within 1 year after receiving study treatment.
* Major surgery within 2 weeks prior to screening, or has surgery scheduled during the study or within 2 weeks after study treatment administration. (Note: Subjects who plan to be conducted surgical procedures under local anesthesia may participate in the study.).
* Any condition which, in the opinion of the investigator, renders the subject unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Within 30 days after cells infusion
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Two years after infusion to the last subject
  The ORR is defined as the percentage of participants who achieve partial response (PR) or better according to international myeloma working group (IMWG) criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China